CLINICAL TRIAL: NCT02912884
Title: Treatment of Polycythaemia Vera and Essential Thrombocythaemia: Influence on the Clot Structure
Acronym: MPNClot
Status: Completed | Type: Observational
Sponsor: Dr Yan Beauverd (Other)
Responsible Party: Sponsor-Investigator, Dr Yan Beauverd, Physician, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: CCER 2016-00950
Record Dates: First submitted 2016-09-10; First posted 2016-09-23 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Polycythemia Vera; Thrombocythemia, Essential
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PV: Patients with a diagnosis of polycythaemia vera.
  Interventions: Drug: No cytoreductive vs cytoreductive drugs
- ET: Patients with a diagnosis of essential thrombocythaemia.
  Interventions: Drug: No cytoreductive vs cytoreductive drugs

INTERVENTIONS:
Drug: No cytoreductive vs cytoreductive drugs — No cytoreductive treatment vs cytoreductive drugs (hydroxycarbamide, alpha-interferon, ruxolitinib).

SUMMARY:
Myeloproliferative neoplasms (MPN) such as Polycythemia Vera (PV) and, Essential Thrombocythaemia (ET) are rare clonal myeloid neoplasms associated with an increased risk of both venous and arterial thrombosis. Thrombotic complications are the main determinant of morbidity and in a less extend mortality.

Routine haemostasis analysis (TP, aPTT) are usually normal and are useless to demonstrate a hypercoagulable state. However, previous evidence suggests that global coagulation tests such as thrombin generation or thromboelastometry are able to detect signs of procoagulant imbalance in MPN. Similarly, current data seems to demonstrate that fibrin clot properties (clot permeability, turbidimetry, clot lysis time) properties is altered suggesting an hypercoagulable state.

Goals of PV and ET treatments are to control blood count to reduce the risk of thrombotic events. Moreover, new drugs such as Janus Kinase Inhibitors (JAKi) were recently licensed for PV and are under investigations on clinical trial for ET. It is currently unknown if treatments that were used for ET and PV, and especially JAKi are able to modify the hypercoagulable state that is observed in those diseases, and if there is difference between drugs.

To evaluate impact of MPN treatment on prothrombotic haemostatic profile, we propose to evaluate global coagulation and fibrin clot properties in MPN, depending on the treatment.

ELIGIBILITY:
Inclusion Criteria:

* All men and women, older than 18 years, with a diagnosis of PV or ET (primary or secondary) according to the 2008 World Health Organization (WHO) classification.

Exclusion Criteria:

* Lack of participant's consent;
* Concomitant treatment with anticoagulant drugs (anti-vitamin K, heparin or direct oral anticoagulant drugs);
* Active cancer other than non-melanoma skin cancer (defined as cancer diagnosis <5 years or treatment <2 years);
* Recent infection (<30d);
* Recent surgery (<30d);
* Recent hospitalization (<30d);
* Recent thromboembolic or cardiovascular event (<3m).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening for participation for MPN patients will occur at the outpatient clinic of the division of Haematology at the Geneva University Hospitals (Rue Gabrielle-Perret-Gentil 4, 1205 Geneva, Switzerland) and at the outpatient clinic of the division of Haematology at Guy's Hospitals (Great Maze Pond, London SE1 9RT, United Kingdom).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Fibrin polymerization; lag-time (in seconds) | At time of inclusion
  Fibrin polymerization will be assessed by turbidity assay on plasma. Fibrin polymerization will be monitored at 340 nm after incubation with human thrombin and CaCl2. Results will report lag-time (seconds).
Fibrin polymerization; maximal absorbance | At time of inclusion
  Fibrin polymerization will be assessed by turbidity assay on plasma. Fibrin polymerization will be monitored at 340 nm after incubation with human thrombin and CaCl2. Results will report maximal absorbance.
Clot lysis time (in minutes) | At time of inclusion
  Fibrinolysis will be assessed by turbidity assay on plasma. Fibrinolysis will be monitored by adding tissue plasminogen activator (tPA). Results will report clot lysis time (minutes)

SECONDARY OUTCOMES:
Clot permeation; permeation coefficient | At time of inclusion
  Clot permeation will be reported as the calculated permeation coefficient (Ks).
Quantitative parameters of thrombin generation test (TGT); endogenous thrombin potential (nM*minutes) | At time of inclusion
  The measurement of thrombin generation is performed by the technique of calibrated automated thrombogram (CAT). Endogenous thrombin potential will be reported in nM*minutes.
Quantitative parameters of thrombin generation test (TGT); peak (nM) | At time of inclusion
  The measurement of thrombin generation is performed by the technique of calibrated automated thrombogram (CAT). Peak will be reported in nM.
Quantitative parameters of thrombin generation test (TGT); time to peak (minutes) | At time of inclusion
  The measurement of thrombin generation is performed by the technique calibrated automated thrombogram (CAT). Time to peak will be reported in minutes.
Fibrin density by laser scanner confocal microscopy (number per 100 μm) | At time of inclusion
  The fibrin density was determined by counting the number of fibres crossing an arbitrary line of 100 μm drawn through a single optical section. Each fibrin clot is prepared in duplicate and 20 density measurements were performed on each sample.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Beauverd, Principal Investigator — University Hospital, Geneva
Locations (2):
- Geneva University Hospitals, Geneva, Switzerland
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No